CLINICAL TRIAL: NCT03171220
Title: Single Center Single Arm Clinical Prospective Study of Neoantigen Reactive T Cells (NRTs) Combined With Programmed Cell Death-1（PD-1） Inhibitor in the Treatment of Chinese Patients With Advanced Refractory Solid Tumors
Brief Title: Neoantigen Reactive T Cells Combined With SHR-1210 for Chinese Patients With Advanced Refractory Solid Tumors
Acronym: NRT-01
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Principal Investigator, Zhengyun Zou, Chief physician, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NDTHNanjing
Record Dates: First submitted 2017-05-13; First posted 2017-05-31 (Actual); Last update posted 2017-06-06 (Actual); Status verified 2017-06

CONDITIONS: Advanced Malignant Solid Tumor
Keywords: Neoantigen; Neoantigen Reactive T cells (NRTs); PD-1 Inhibitor; Advanced Solid Tumor; Adoptive Cell Therapy(ACT); PD-1 antibody; SHR1210
MeSH Terms: interventions — camrelizumab; fludarabine; Cyclophosphamide; Interleukin-2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neoantigen Reactive T Cells + SHR-1210 (Experimental): Peripheral blood lymphocytes will be collected and neoantigen reactive T cells(NRTs) will be generated in the laboratory;Both Fludarabine 30mg/m2/D and Cyclophosphamide 300mg/m2/D will be i.v. for 3 days before cell infusion; NRTs 0.5~1 x 10^10, will be i.v.Q3 weeks for total 4 doses;programmed cell death-1（PD1） inhibitor SHR-1210,200mg,will be i.v. Q3 weeks for total 4 doses,2 day2 prior to each NRTs infusion;Interleukin-2 (IL-2) will be continuous intravenous infused since the first day of the cell infusion for 5 consecutive days, 4000,000 international unit per day.All Patients will receive a total of 4 cycles of treatment.
  Interventions: Biological: Neoantigen Reactive T Cells(NRTs); Biological: SHR-1210; Drug: Fludarabine; Drug: Cyclophosphamide; Biological: Interleukin-2

INTERVENTIONS:
Biological: Neoantigen Reactive T Cells(NRTs) — Neoantigen Reactive T Cells in an expected volume of 100 milliliter（mL） will be given by intravenous injection over 2-10 minutes through either a peripheral or a central line.
Biological: SHR-1210 — SHR-1210 200mg will be administered as an intravenous infusion over 60 minutes.
Drug: Fludarabine — Fludarabine(FLU) 30mg/m2/d×3d，3 days prior to each NRTs infusion as preconditional chemotherapy.
  Other Names: FLU
Drug: Cyclophosphamide — Cyclophosphamide(CTX) 300mg/m2/d×3d，3 days prior to each NRTs infusion as preconditional chemotherapy.
  Other Names: CTX
Biological: Interleukin-2 — Interleukin-2(IL-2)will be continuous intravenous infused since the first day of the cell infusion for 5 consecutive days, 4000,000 international unit per day.
  Other Names: IL-2

SUMMARY:
The purpose of this study is to see the safety and efficient of neoantigen reactive T cells (NRTs) combined with programmed cell death-1(PD-1) inhibitor（SHR-1210）in the treatment of Chinese patients with advanced refractory solid tumors.

DETAILED DESCRIPTION:
The tumor-specific "none-self" immunogenic neoantigens encoded by either viral genes or somatic mutation genes, possess the potential to induce specific anti-cancer immunity, including cellular and humoral immune responses. Today, numerous clinical trials demonstrate that although these "none-self" antigens initiate the antigen-specific immunoglobulin G antibodies and cluster of differentiation 4（CD4）+/cluster of differentiation 8（CD8）+T-cells response, not all of them show a clinical benefit in the response rate, progression-free survival or overall survival.Immune tolerance induced by PD-1 or programmed cell death-ligand1（ PD-L1）maybe play a vital role for these negative outcomes.Personalized cell therapy plus checkpoint inhibitors maybe own a breakthrough in the treatment of those malignant diseases without standard options.Our center has successfully established a new method for preparing personalized neoantigen reactive T cells(NRTS) for adoptive cell therapy(ACT). Today, we will carry out a single center single arm clinical prospective study of NRTs combined with PD-1 inhibitor(SHR-1210) for the treatment of Chinese patients with advanced refractory solid tumors. Participants are assigned to receive 4 circles of cell therapy,and prior to each cycle's immunocytes treatment,preconditional chemotherapy and SHR-1210 will be carried out, and IL-2 continuous intravenous infusion（CIV） will also be given for 5 consecutive days after each time's cell infusion. The safety and clinical response rate（RR） are evaluated. Biomarkers and immunological markers are also monitored.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 18 to 75 years old
* Histologic or cytologic confirmation of advanced refractory solid tumors with no available curative treatment options
* At least one measurable disease: diameter ≥20mm or spiral computed tomography(CT)≥10mm; and can providing with tumor specimen (for testing the expression of PD -L1 and the infiltrating lymphocytes)
* Must be human leukocyte antigen (HLA)-A2/A24/A11 positive
* Eastern Cooperative Oncology Group(ECOG)<0-2 and expected survival time 3 months or more
* At least one new antigen can induce T cell secrete interferon - gamma (IFN - gamma) twice as normal controls during the new antigens screening
* Without anticancer treatment more than one month
* Hematology Index including: Neutrophile granulocyte greater than 1.5×10^9/L; Hemoglobin greater than 10g/dL; Platelet greater than 100×10^9/L
* Biochemical index including: Serum bilirubin not greater than 1.5x upper limit of reference range (ULN); glutamic-pyruvic transaminase（ALT） or glutamic-oxalacetic transaminase（AST） not greater than 2.5x ULN; Creatinine clearance no less than 60ml/min
* Peripheral venous channel open and no contraindications to separating lymphocytes
* Negative pregnancy test for women of childbearing potential, and patients must be willing to practice birth control during the regimen
* Provision of informed consent
* Be able to follow the research program and follow up process

Exclusion Criteria:

* Those who now are undergoing other antitumor drug therapy (including chemotherapy, systemic steroids therapy, surgery, target therapy or immune therapy);
* Prior treatment with PD-1 monoclonal antibody(mAb） or PD-L1 mAb;
* Prior malignancy active within the previous 5 years except for locally curable cancers that have been apparently cured, such as basal cell skin cancer or carcinoma in situ of the cervix;
* History with pulmonary tuberculosis, and positive tests for Acquired Immune Deficiency Syndrome(HIV),hepatitis C virus(HCV),hepatitis B virus(HBV);
* Patients with any active autoimmune disease or a documented history of autoimmune disease, or history of syndrome that required systemic steroids or immunosuppressive medications, such as hypophysitis, pneumonia, colitis, hepatitis, nephritis, hyperthyroidism or hypothyroidism; Severe, uncontrolled medical condition that would affect patients' compliance or obscure the interpretation of toxicity determination or adverse events, including active severe infection, uncontrolled diabetes, angiocardiopathy (heart failure > class II New York Heart Association(NYHA), heart block >II grade, myocardial infarction, unstable arrhythmia or unstable angina within past 6 months, cerebral infarction within past 3 months) or pulmonary disease ( interstitial pneumonia, obstructive pulmonary disease or symptomatic bronchospasm).
* Evidence with central nervous system(CNS) disease
* Pregnant or nursing
* Psychiatric medicines abuse without withdrawal, or history of psychiatric illness.
* Hypersensitivity to investigational drugs or its components.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-06-01 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Adverse Events | up to 6 months
  using Common Terminology Criteria for Adverse Events (CTCAE v4.0) in patients

SECONDARY OUTCOMES:
Response Rate | At 3, 6 and 12 months
  Response Rate（RR） will be evaluated according Response Evaluation Criteria in Solid Tumors
Progression free survival (PFS) | At 6,9 and 12 months
  the duration of progression free survival is measured from the time of treatment to the first date that recurrent or progressive disease or for any reason of death is objectively documented.

OTHER OUTCOMES:
Overall Survival (OS) | At 6,12 and 18 months
  the duration is measured from the time of treatment to the time of death
Interferon-gama change of PBMC cells in the peripheral blood stimulated by tumor antigens | At baseline,40days,2 months,6 months and at the time of disease progress
  T cells in the peripheral blood stimulated by tumor antigens for 24 hr，and then Interferon-gama secretion is measured
Th1/Th2 change in the peripheral blood | At baseline,40days,2 months,6 months and at the time of disease progress
  cytokines are measured by flow cytometry(FCM)

CONTACTS AND LOCATIONS:
Overall Officials: Baorui Liu, M.D & Ph.D, Principal Investigator — The Comprehensive Cancer Centre of Nanjing Drum Tower Hospital
Locations (1):
- The Comprehensive Cancer Centre of Drum Tower Hospital, Medical School of Nanjing University and Clinical Cancer Institute of Nanjing University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Gros A, Parkhurst MR, Tran E, Pasetto A, Robbins PF, Ilyas S, Prickett TD, Gartner JJ, Crystal JS, Roberts IM, Trebska-McGowan K, Wunderlich JR, Yang JC, Rosenberg SA. Prospective identification of neoantigen-specific lymphocytes in the peripheral blood of melanoma patients. Nat Med. 2016 Apr;22(4):433-8. doi: 10.1038/nm.4051. Epub 2016 Feb 22. PMID 26901407
- [Result] Desrichard A, Snyder A, Chan TA. Cancer Neoantigens and Applications for Immunotherapy. Clin Cancer Res. 2016 Feb 15;22(4):807-12. doi: 10.1158/1078-0432.CCR-14-3175. Epub 2015 Oct 29. PMID 26515495
- [Result] Rosenberg SA, Restifo NP. Adoptive cell transfer as personalized immunotherapy for human cancer. Science. 2015 Apr 3;348(6230):62-8. doi: 10.1126/science.aaa4967. PMID 25838374
- [Result] Su S, Zou Z, Chen F, Ding N, Du J, Shao J, Li L, Fu Y, Hu B, Yang Y, Sha H, Meng F, Wei J, Huang X, Liu B. CRISPR-Cas9-mediated disruption of PD-1 on human T cells for adoptive cellular therapies of EBV positive gastric cancer. Oncoimmunology. 2016 Nov 22;6(1):e1249558. doi: 10.1080/2162402X.2016.1249558. eCollection 2017. PMID 28197365
- [Result] Stevanovic S, Pasetto A, Helman SR, Gartner JJ, Prickett TD, Howie B, Robins HS, Robbins PF, Klebanoff CA, Rosenberg SA, Hinrichs CS. Landscape of immunogenic tumor antigens in successful immunotherapy of virally induced epithelial cancer. Science. 2017 Apr 14;356(6334):200-205. doi: 10.1126/science.aak9510. PMID 28408606
- [Result] Tran E, Robbins PF, Lu YC, Prickett TD, Gartner JJ, Jia L, Pasetto A, Zheng Z, Ray S, Groh EM, Kriley IR, Rosenberg SA. T-Cell Transfer Therapy Targeting Mutant KRAS in Cancer. N Engl J Med. 2016 Dec 8;375(23):2255-2262. doi: 10.1056/NEJMoa1609279. PMID 27959684
- [Result] Parkhurst M, Gros A, Pasetto A, Prickett T, Crystal JS, Robbins P, Rosenberg SA. Isolation of T-Cell Receptors Specifically Reactive with Mutated Tumor-Associated Antigens from Tumor-Infiltrating Lymphocytes Based on CD137 Expression. Clin Cancer Res. 2017 May 15;23(10):2491-2505. doi: 10.1158/1078-0432.CCR-16-2680. Epub 2016 Nov 8. PMID 27827318
- [Derived] Chen F, Zou Z, Du J, Su S, Shao J, Meng F, Yang J, Xu Q, Ding N, Yang Y, Liu Q, Wang Q, Sun Z, Zhou S, Du S, Wei J, Liu B. Neoantigen identification strategies enable personalized immunotherapy in refractory solid tumors. J Clin Invest. 2019 Mar 5;129(5):2056-2070. doi: 10.1172/JCI99538. Print 2019 May 1. PMID 30835255